CLINICAL TRIAL: NCT02983968
Title: Use of the French Healthcare Insurance Database to Evaluate How Early Diagnosis of Hepatocellular Carcinomas is Implemented in France: SAMHEPAT Study
Brief Title: Use of the French Healthcare Insurance Database
Acronym: SAMHEPAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2015-43 Pr Ganry
Record Dates: First submitted 2016-11-30; First posted 2016-12-06 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Cirrhosis
Keywords: Oncology; Hepatology; Public Health; Liver
MeSH Terms: conditions — Fibrosis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Other: Description of the cirrhosis management

SUMMARY:
Hepatocellular carcinoma (HCC) has become the second most common cause of cancer death in the world, estimated responsible for nearly 745,000 deaths in 2012 (9.1% of all cancer deaths).

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) has become the second most common cause of cancer death in the world, estimated responsible for nearly 745,000 deaths in 2012 (9.1% of all cancer deaths). This cancer is closely associated with the presence of chronic liver underlying disease and early diagnosis following a systematic surveillance of cirrhotic patients could improve disease-free survival in patients declaring HCC. However, the risk-benefit ratio of such monitoring is discussed. Nevertheless, it is recommended in patients with liver cirrhosis, from which the prevalence is estimated between 0.3% and 0.6% in the French population. This debate can lead to a failure to comply with recommendations and promote a large variability in the management of the surveillance of HCC in patients with cirrhosis in practice. Data acquisition regarding the current situation in France is required.

The objective of this project is to use this database to document current practices concerning monitoring of incidents HCC in cirrhotic patients in France. A retrospective cohort study will be conducted on data from SNIIRAM recorded between 2007 and 2015. The primary analysis will focus on multivariate modelling of the deviation rate from the recommendations (advising the realisation of at least two echodoppler ultrasonographies yearly) with a competitive risk model, taking into account gender, social status, Charlson index, age at baseline, the alcoholic etiology of cirrhosis, type of facility and the yearly number of visits to a hepatologist during follow-up. It is estimated that more than 86,000 patients with a minimum follow-up of 3 years will be included in the analysis

ELIGIBILITY:
Inclusion Criteria:

- Cirrhotic patients aged between 18 and 75 years.

(A cirrhotic patient will be defined as a presenting a first occurrence of a codes used in hospitalisation for cirrhosis or as a motive for granting an ALD 6 (cirrhosis motivated) financial support )

Exclusion Criteria:

- None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic patients aged between 18 and 75 years
Sampling Method: Non-Probability Sample
Enrollment: 890 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Rate of deviation from the guidelines | 01/01/2007 - 01/01/2018

SECONDARY OUTCOMES:
Factors associated with deviation from the guidelines | 01/01/2007 - 01/01/2018
  A multivariate regression analysis will be performed to objectivate factors associated with the deviation among sex, poor social status, Charlson index, age at inclusion and the alcoholic aetiology of the cirrhosis, type facility where hospitalisation occurred, number of hepatologist visits and living area

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GANRY, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France